CLINICAL TRIAL: NCT06819020
Title: Adaptive Deep Brain Stimulation to Improve Freezing of Gait in Parkinson's Disease Using Percept RC
Brief Title: Adaptive Deep Brain Stimulation for Freezing of Gait in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Doris Wang, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Doris Wang, MD, PhD, Associate Professor, Neurological Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25-43493
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Neuromodulation; Deep Brain Stimulation; Freezing of Gait; Adaptive DBS; Gait Impairment; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: In a small, double-blinded trial, the investigators will compare the effects of aDBS versus conventional open-loop DBS on gait. Participants will be randomized to either open-loop DBS or different aDBS conditions (10 days per condition, with counterbalancing the order of stimulation within subject and randomizing this counterbalanced order across subjects). Participants will be perform gait tasks at home along with doing their everyday activities with a wearable device that tracks gait metrics and FOG episodes. Gait and balance measurements, external wearable data collection, and UPDRS III will be performed at the end of the 10-day stimulation period for each condition in-person.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Open-loop deep brain stimulation (Active Comparator): Participants with Parkinson's disease implanted with Percept RC and brain lead implanted in the pallidal/striatal region receiving open-loop deep brain stimulation.
  Interventions: Device: Percept RC
- Adaptive deep brain stimulation (ramp-up) (Active Comparator): Participants with Parkinson's disease implanted with Percept RC and brain lead implanted in the pallidal/striatal region receiving increased stimulation in-response to gait-behavior biomarker.
  Interventions: Device: Percept RC
- Adaptive deep brain stimulation (ramp-down) (Active Comparator): Participants with Parkinson's disease implanted with Percept RC and brain lead implanted in the pallidal/striatal region receiving decreased stimulation in-response to gait-behavior biomarker.
  Interventions: Device: Percept RC

INTERVENTIONS:
Device: Percept RC — Using the Percept RC pulse generator, patients receive clinically-optimized open loop stimulation to the pallidum/subthalmaic nucleus.
  Other Names: Continuous deep brain stimulation
  Arms: Open-loop deep brain stimulation
Device: Percept RC — Using the Percept RC pulse generator, patients receive increased adaptive stimulation to the pallidum/subthalmaic nucleus.
  Other Names: Adaptive deep brain stimulation
  Arms: Adaptive deep brain stimulation (ramp-up)
Device: Percept RC — Using the Percept RC pulse generator, patients receive decreased adaptive stimulation to the pallidum/subthalmaic nucleus.
  Other Names: Adaptive deep brain stimulation
  Arms: Adaptive deep brain stimulation (ramp-down)

SUMMARY:
The goal of this clinical trial is to learn if adaptive deep brain stimulation (DBS) can decrease or prevent freezing of gait in participants with Parkinson's disease.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. Does adaptive DBS lead to fewer freezing of gait episodes for participants compared to their clinical continuous DBS settings?
2. Does adaptive DBS change other parts of participants' walking, like step length, step time, or step symmetry?

Investigators will compare personalized adaptive DBS settings for each participant with their continuous DBS settings to see if adaptive DBS works better to treat gait symptoms, including freezing of gait.

Participants will have DBS insertion surgery as part of their standard medical care. Along with the DBS system, they will also have permanent sensors placed between their skull and scalp to detect brain activity related to movement. After, participants will:

1. Measure their walking using at-home monitoring devices (worn on the hip or ankles) while on their clinical continuous DBS settings.
2. Visit the lab for check-ins and testing of adaptive DBS settings.
3. Try different adaptive DBS settings at home, while wearing at-home monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent for the study
2. Movement disorder symptoms that are sufficiently severe, in spite of best medical therapy, to warrant surgical implantation of deep brain stimulators according to standard clinical criteria
3. Patient has requested surgical intervention with deep brain stimulation for their disorder
4. No magnetic resonance (MR) abnormalities that suggest an alternative diagnosis or contraindicate surgery
5. Absence of significant cognitive impairment (score of 21 or greater on the Montreal Cognitive Assessment (MoCA)),
6. Signed informed consent
7. Ability to comply with study follow-up visits for brain recording, testing of adaptive stimulation, and clinical assessment.
8. Age 21-75
9. Diagnosis of idiopathic PD with duration of motor symptoms for 3 years or greater
10. Patient has undergone appropriate therapy with oral medications with inadequate relief as determined by a movement disorders neurologist.
11. UPDRS-III score off medication between 20 and 80 and an improvement of at least 30% in the baseline UPDRS-III on medication score, compared to the baseline off-medication score, and motor fluctuations with at least 2 hours per day of on time without dyskinesia or with non-bothersome dyskinesia.

    OR Patients with tremor-dominant PD (a tremor score of at least 2 on a UPDRS-III sub-score for tremor), treatment resistant, with significant functional disability despite maximal medical management
12. Patients with gait impairments including freezing of gait off medication.
13. Ability of patient and/or caregivers to recharge the system evaluated by all clinicians and study personnel.

Exclusion Criteria:

1. Coagulopathy, anticoagulant medications, uncontrolled hypertension, history of seizures, heart disease, or other medical conditions considered to place the patient at elevated risk for surgical complications
2. Evidence of a psychogenic movement disorder: Motor symptoms that remit with suggestion or "while unobserved", symptoms that are inconsistent over time or incongruent with clinical condition, plus other manifestation such as "false" signs, multiple somatizations, or obvious psychiatric disturbance.
3. Pregnancy: all women of child bearing potential will have a negative urine pregnancy test prior to undergoing their surgical procedure.
4. Significant untreated depression (BDI-II score >20). History of suicidal attempt or active suicidal ideation (Yes to #2-5 on C-SSRS)
5. Any personality or mood symptoms that study personnel believe will interfere with study requirements.
6. Subjects who require Electroconvulsive therapy (ECT), Repetitive Transcranial Magnetic Stimulation (rTMS) or diathermy
7. Implanted stimulation systems such as cochlear implant, pacemaker, defibrillator, or neurostimulator
8. Previous cranial surgery
9. Drug or alcohol abuse
10. Meets criteria for Parkinson's disease with mild cognitive impairment (PD-MCI). These criteria are performance of more than two standard deviations below appropriate norms, for tests from two or more of these five cognitive domains: attention, executive function, language, memory, and visuospatial tests.
11. Known allergies to the implantable device components including titanium, polyurethane, silicone, and nylon.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Freezing of gait | Baseline and 2 years
  Freezing of gait episodes will be detected using validated home wearable devices along with participant self-reporting.

SECONDARY OUTCOMES:
Change in Gait | Baseline and 2 years
  Change in gait measurements using the 10-meter walk timed test. The 10-Meter Walk Test (10MWT) is a performance measure used to assess walking speed in meters per second over a short distance of 10 meters. It is employed to determine functional mobility and gait. The gait speed is used as the outcome by which to compare change in performance capacity. Lower times indicate higher levels of physical functioning.
Change in Balance | Baseline and 2 years
  Change in balance measurements using:
  Mini-BESTest Clinical balance assessment tool. The score range is 0-2 with high score indicating higher levels of physical functioning.
Change in MDS-UPDRS III scores | Baseline and 2 years
  Change in Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) III score. The scale consists of 18 items that are each scored 0 to 3, making the total score out of 72 points, with higher scores indicating higher impairment.
Change in Stride Length | Baseline and 2 years
  Change in stride length measured by Rover (a gait measurement device), Xsens (a kinematic measurement device), and Stat-On (a gait measurement device), with adaptive compared to open-loop deep brain stimulation (DBS). Stride length is measured in meters.
Change in Stride Time | Baseline and 2 years
  Change in stride time measured by Rover (a gait measurement device), Xsens (a kinematic measurement device), and Stat-On (a gait measurement device) with adaptive compared to open-loop deep brain stimulation (DBS). Stride time is measured in seconds.
Change in Arm Swing Amplitude | Baseline and 2 years
  Change in arm swing ampliture measured Xsens (a kinematic measurement device) with adaptive compared to open-loop deep brain stimulation (DBS). Arm swing amplitude is measured in meters.
Change in Gait Symmetry | Baseline and 2 years
  Change in gait symmetry measured by Rover (a gait measurement device), Xsens (a kinematic measurement device), and Stat-On (a gait measurement device), with adaptive compared to open-loop deep brain stimulation (DBS).
Change in Gait Variance | Baseline and 2 years
  Change in gait variance measured by Rover (a gait measurement device), Xsens (a kinematic measurement device), and Stat-On (a gait measurement device), with adaptive compared to open-loop deep brain stimulation (DBS).
Change in Total Electrical Energy Delivered (TEED) | Baseline and 2 years
  Change in TEED calculated using voltage, frequency, pulse width, and impedence values from participant pulse generators, with adaptive compared to open-loop deep brain stimulation (DBS). TEED is measured in microjoules.

CONTACTS AND LOCATIONS:
Overall Officials: Doris D Wang, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No